CLINICAL TRIAL: NCT03052517
Title: A 2-treatment Period, Randomized, Placebo-controlled, Multicenter Parallel-group Study to Assess the Safety of QAW039 When Added to Existing Asthma Therapy in GINA Steps 3, 4 and 5 Patients With Uncontrolled Asthma.
Brief Title: Study of Safety of QAW039 in Patients With Asthma Inadequately Controlled on Standard-of-care Asthma Treatment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAW039A2315; 2016-001560-11 (EudraCT Number)
Record Dates: First submitted 2017-01-23; First posted 2017-02-14 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Asthma
Keywords: Asthma; QAW039; allergic asthma; allergy triggered asthma; reactive asthma; asthma attack; difficulty breathing
MeSH Terms: conditions — Asthma; Dyspnea | interventions — fevipiprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- QAW039 150mg (Experimental): QAW039 Dose 1 once daily
  Interventions: Drug: QAW039 150 mg
- QAW039 450 mg (Experimental): QAW039 Dose 2 once daily
  Interventions: Drug: QAW039 450 mg
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAW039 150 mg — One tablet of QAW039 150 mg once daily
  Arms: QAW039 150mg
Drug: QAW039 450 mg — One tablet of QAW039 450 mg once daily
  Arms: QAW039 450 mg
Drug: Placebo — One tablet of Placebo once daily
  Arms: Placebo

SUMMARY:
This study was a 2-treatment period, randomized, multicenter parallel-group study. The overall purpose of this study was to provide long- term safety data for fevipiprant (QAW039) (Dose 1 and Dose 2), compared with placebo, when added to the Global Initiative for Asthma (GINA) steps 3, 4, and 5 standard-of-care (SoC) asthma therapy (GINA 2016), in patients with moderate-to- severe asthma.

The purpose of this study was to provide long-term safety data for QAW039 150 mg once daily and 450 mg once daily, compared with placebo, when added to GINA steps 3, 4, and 5 standard-of-care asthma therapy (GINA 2020) in adult and adolescent (≥12 years) patients with moderate-to-severe asthma. The study included 2 cohorts of patients:

1. Rollover patients who had completed any of the four Phase 3 pivotal efficacy studies with QAW039 (QAW039A2307, QAW039A2314, QAW039A2316, or QAW039A2317, hereafter referred to as Studies A2307, A2314, A2316, and A2317), thus providing data for a longer duration of exposure, and
2. New patients who had not previously participated in a study of QAW039, permitting an increase in the number of patients with long-term exposure to QAW039.

By including these 2 categories of patients, the total number of patients treated with QAW039 as well as the duration of exposure to QAW039 treatment was substantially increased, supporting evaluation of the safety profile of QAW039.

DETAILED DESCRIPTION:
The study comprised 2-treatment period. Treatment Period 1 was a 52-week, double-blind treatment period in which QAW039 450 mg or 150 mg or placebo was added to standard-of-care asthma therapy according to GINA guidelines. Treatment Period 2 was an optional 104-week, single-blind treatment period in which patients received QAW039 450 mg or 150 mg or placebo added to standard-of-care asthma therapy according to GINA guidelines.

ELIGIBILITY:
Inclusion Criteria:

Patients completing a prior Phase 3 study of QAW039:

* Informed consent and assent (if applicable).
* Completion of the Treatment Period (on blinded study drug) of a prior Phase 3 study of QAW039.
* Patient is able to safely continue into the study as judged by the investigator.

Patients who have not previously participated in a study of QAW039:

* Written informed consent.
* A diagnosis of asthma,uncontrolled on GINA 3/4/5 asthma medication.
* Evidence of airway reversibility or airway hyper- reactivity.
* FEV1 of ≤85% of the predicted normal value.
* An ACQ score ≥1.5 prior to entering the study.

Exclusion Criteria:

Patients completing a prior phase 3 study of QAW039:

* Pregnant or nursing (lactating) women.
* Women of child-bearing potential unless they are using basic methods of contraception during dosing of study drug
* Patients who did not complete the Treatment Period on blinded study drug of the prior QAW039 study they participated in.
* Inability to comply with all study requirements.
* Patient who experienced a serious and drug-related AE in the prior QAW039 study they participated in.

Patients who have not previously participated in a study of QAW039:

* Use of other investigational drugs within 5 half-lives of study entry, or within 30 days, whichever is longer.
* Subjects who have participated in another trial of QAW039 (i.e.-the patient was randomized in another study).
* A QTcF (Fridericia) ≥450 msec (male) or ≥460 msec (female).
* History of malignancy with the exception of local basal cell carcinoma of the skin
* Pregnant or nursing (lactating) women.
* Serious co-morbidities.
* Patients on greater than 20 mg of simvastatin> 40 mg of atorvastatin, >40 mg of pravastatin, or >2 mg of pitavastatin. Statin doses less than or equal to these doses as well as other statins will be permitted during the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2538 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (296):
- United States (44):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Encinitas, California
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Westminster, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Lafayette, Colorado
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Zachary, Louisiana
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Waldorf, Maryland
  - Novartis Investigative Site, Ypsilanti, Michigan
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigative Site, Bellevue, Nebraska
  - Novartis Investigative Site, La Vista, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Gastonia, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Edmond, Oklahoma
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Altoona, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, East Providence, Rhode Island
  - Novartis Investigative Site, Boerne, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Bellingham, Washington
  - Novartis Investigative Site, Spokane, Washington
- Argentina (14):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Ranelagh, Partido de Berazate, Buenos Aires
  - Novartis Investigative Site, Santa Rosa, La Pampa Province
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Salta
  - Novartis Investigative Site, Santa Fe
- Australia (3):
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Footscray, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
- Austria (2):
  - Novartis Investigative Site, Feldkirch
  - Novartis Investigative Site, Vienna
- Belgium (7):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Erpent
  - Novartis Investigative Site, Éghezée
  - Novartis Investigative Site, Herentals
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Liège
- Brazil (8):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Porto Alegre, Porto Alegre RS
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, São Bernardo do Campo, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Sorocaba, São Paulo
- Bulgaria (4):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
- Canada (6):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec
  - Novartis Investigative Site, Vancouver
- China (10):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
- Colombia (3):
  - Novartis Investigative Site, Ibagué, Tolima Department
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Bucaramanga
- Czechia (6):
  - Novartis Investigative Site, Jindřichův Hradec, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Teplice, CZE
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Karlovy Vary
  - Novartis Investigative Site, Mladá Boleslav
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Novartis Investigative Site, Helsinki, Finland
- France (8):
  - Novartis Investigative Site, Montpellier, Herault
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
- Germany (7):
  - Novartis Investigative Site, Cottbus, Saxony
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Landsberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Witten
- Greece (3):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Guatemala (3):
  - Novartis Investigative Site, Gautemala City, Gautemala
  - Novartis Investigative Site, Guatemala City, GTM
  - Novartis Investigative Site, Guatemala City
- Hungary (13):
  - Novartis Investigative Site, Budaörs, HUN
  - Novartis Investigative Site, Győr, HUN
  - Novartis Investigative Site, Hajdúnánás, HUN
  - Novartis Investigative Site, Püspökladány, HUN
  - Novartis Investigative Site, Százhalombatta, HUN
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Komárom
  - Novartis Investigative Site, Makó
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Siófok
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Törökbálint
- India (8):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Dehradun, Uttarakhand
- Israel (5):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
- Japan (38):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Chikushino-shi, Fukuoka
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Kasuga, Fukuoka
  - Novartis Investigative Site, Koga, Fukuoka
  - Novartis Investigative Site, Yanagawa, Fukuoka
  - Novartis Investigative Site, Mizunami, Gifu
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Naka-gun, Ibaraki
  - Novartis Investigative Site, Sakaidechō, Kagawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kōshi, Kumamoto
  - Novartis Investigative Site, Matsusaka, Mie-ken
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Habikino, Osaka
  - Novartis Investigative Site, Kishiwada, Osaka
  - Novartis Investigative Site, Tokyo, Shibuya Ku
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Setagaya-Ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Toshima Ku, Tokyo
- Latvia (2):
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Lebanon (3):
  - Novartis Investigative Site, El Chouf, LBN
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
- Lithuania (5):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius, LTU
  - Novartis Investigative Site, Kaunas, LT
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Vilnius
- Malaysia (3):
  - Novartis Investigative Site, Kota Bharu, Kelantan
  - Novartis Investigative Site, Kuantan, Pahang
  - Novartis Investigative Site, Taiping, Perak
- Mexico (3):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Guadalajara Jalisco, Jalisco
  - Novartis Investigative Site, Río de Janeiro
- Netherlands (2):
  - Novartis Investigative Site, Arnhem
  - Novartis Investigative Site, Leeuwarden
- Peru (6):
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Martín de Porres, Lima region
  - Novartis Investigative Site, Cusco
  - Novartis Investigative Site, Lima
  - Novartis Investigative Site, Piura
- Philippines (6):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Quezon City, Manila
  - Novartis Investigative Site, Bulacan
  - Novartis Investigative Site, Iloilo City
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
- Poland (4):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Strzelce Opolskie
- Novartis Investigative Site, San Juan, Puerto Rico
- Romania (7):
  - Novartis Investigative Site, Bucharest, District 3
  - Novartis Investigative Site, Constanța, ROM
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Bragadiru
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Deva
- Russia (14):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Stavropol
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Jeddah, Saudi Arabia
- Serbia (4):
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Kamenitz
  - Novartis Investigative Site, Kragujevac
  - Novartis Investigative Site, Niš
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (10):
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Kežmarok
  - Novartis Investigative Site, Komárno
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Spišská Nová Ves
  - Novartis Investigative Site, Žilina
- Spain (14):
  - Novartis Investigative Site, Marbella, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Jerez de la Frontera, Cadiz
  - Novartis Investigative Site, Laredo, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Barcelona, Vic
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, Guadalajara
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Santiago de Compostela
  - Novartis Investigative Site, Zaragoza
- Switzerland (2):
  - Novartis Investigative Site, Liestal
  - Novartis Investigative Site, Lugano
- Novartis Investigative Site, Taichung, Taiwan
- Turkey (Türkiye) (6):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Bursa
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Yenisehir/Izmir
- United Kingdom (6):
  - Novartis Investigative Site, Cambridge, Cambrigdeshire
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, Chertsey, Surrey
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, Leicester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Maspero J, Agache IO, Kamei T, Yoshida M, Boone B, Felser JM, Kawakami F, Knorr B, Lawrence D, Lehmann T, Wang W, Pedinoff AJ. Long-term safety and exploratory efficacy of fevipiprant in patients with inadequately controlled asthma: the SPIRIT randomised clinical trial. Respir Res. 2021 Dec 11;22(1):311. doi: 10.1186/s12931-021-01904-8. PMID 34895218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were from ARG, AUS, AUT, BEL, BRA, BGR, CAN, CHN, COL, CZE, EST, FIN, FRA, DEU, GRC, GTM, HUN, IND, ISR, JPN, LVA, LBN, LTU, MYS, MEX, NLD, PER, PHL, POL, ROU, RUS, SAU, SRB, SGP, SVK, ESP, CHE, TWN, TUR, GBR, USA
Pre-assignment Details: Eligible patients included patients completing a prior QAW039 Phase 3 study (CQAW039A2307, QAW039A2314, CQAW039A2316, or CQAW039A2317) and patients who had not previously participated in a QAW039 study.
Period: Overall Study
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Started | 1093 | 1085 | 360
Safety Set (SAF) (All patients who received at least one dose of study drug during this study.) | 1092 (One patient received placebo. This patient was not included in QAW039 150 mg group in the SAF) | 1084 (One patient had no treatment administered and thus was excluded from the SAF) | 361 (One patient in QAW039 150 mg group received placebo and was included in the placebo group in the SAF)
Completed | 76 | 71 | 32
Not Completed | 1017 | 1014 | 328
Not completed — Study Terminated By Sponsor | 928 | 938 | 296
Not completed — Subject/Guardian Decision | 50 | 45 | 22
Not completed — Lack of Efficacy | 23 | 14 | 7
Not completed — Adverse Event | 6 | 5 | 0
Not completed — Physician Decision | 4 | 5 | 1
Not completed — Death | 3 | 0 | 1
Not completed — Lost to Follow-up | 2 | 4 | 0
Not completed — Pregnancy | 1 | 0 | 1
Not completed — Non-Compliance With Study Treatment | 0 | 2 | 0
Not completed — Technical Problems | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: SAF: All patients who received at least one dose of study drug during this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo | Total
Number analyzed (Participants) | 1092 | 1084 | 361 | 2537
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.1 (14.95) | 50.1 (15.55) | 49.9 (14.99) | 50.1 (15.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 659 | 666 | 229 | 1554
  Male | 433 | 418 | 132 | 983
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 757 | 756 | 243 | 1756
  Black | 30 | 14 | 11 | 55
  Asian | 219 | 215 | 73 | 507
  Native American | 27 | 40 | 12 | 79
  Pacific Islander | 0 | 1 | 0 | 1
  Unknown | 0 | 9 | 2 | 11
  Other | 59 | 49 | 20 | 128

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) up to Week 52 - Cox Regression Model
Description: Adverse events starting on or after the day of the first intake of study drug in this study and until the day of last intake of study drug +7 days (30 days in the case of a serious AE) were classified as treatment emergent AEs. For this Outcome Measure, AE up to week 52 are reported.
Time Frame: 52 weeks
Population: Safety analysis set (SAF): included all patients who received at least one dose of study drug during this study. Patients were analyzed according to the treatment they received during this study. Only patients with data for all terms in the Cox regression model were included
Measure: Count of Participants; unit: Participants
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 1081 | 1077 | 359
Participants | 675 | 654 | 237
Statistical Analysis 1: Comparison: QAW039 150mg vs Placebo; Hazard Ratio = QAW039 150mg / Placebo; Test type: Other; Regression, Cox; The Cox regression model = treatment group+ severity of asthma + region as fixed class effects, stratified by randomization stratum; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.74 to 1.00] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Hazard Ratio = QAW039 450mg / Placebo; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.72 to 0.97] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio
Statistical Analysis 3: Comparison: QAW039 150mg vs QAW039 450 mg; Hazard Ratio = QAW039 450mg / QAW039 150mg; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.87 to 1.09] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) up to Week 156 - Cox Regression Model
Description: Adverse events starting on or after the day of the first intake of study drug in this study and until the day of last intake of study drug +7 days (30 days in the case of a serious AE) were classified as treatment emergent AEs
Time Frame: 156 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 1081 | 1077 | 359
Participants | 709 | 681 | 243
Statistical Analysis 1: Comparison: QAW039 150mg vs Placebo; Hazard Ratio = QAW039 150mg / Placebo; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.76 to 1.02] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Hazard Ratio = QAW039 450mg / Placebo; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.73 to 0.99] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio
Statistical Analysis 3: Comparison: QAW039 150mg vs QAW039 450 mg; Hazard Ratio = QAW039 450mg / QAW039 150mg; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.86 to 1.08] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio

3. Primary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (SAEs) up to Week 52 - Cox Regression Model
Description: Serious Adverse events starting on or after the day of the first intake of study drug in this study and until the day of last intake of study drug +30 days were classified as treatment emergent SAEs. For this Outcome Measure, AE up to week 52 are reported.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 1081 | 1077 | 359
Participants | 73 | 53 | 29
Statistical Analysis 1: Comparison: QAW039 150mg vs Placebo; Hazard Ratio = QAW039 150mg / Placebo; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.51 to 1.22] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Hazard Ratio = QAW039 450mg / Placebo; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.39 to 0.97] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio
Statistical Analysis 3: Comparison: QAW039 150mg vs QAW039 450 mg; Hazard Ratio = QAW039 450mg / QAW039 150mg; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.54 to 1.14] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio

4. Primary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (SAEs) up to Week 156 - Cox Regression Model
Description: Serious Adverse events starting on or after the day of the first intake of study drug in this study and until the day of last intake of study drug +30 days were classified as treatment emergent SAEs.
Time Frame: 156 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 1081 | 1077 | 359
Participants | 86 | 63 | 33
Statistical Analysis 1: Comparison: QAW039 150mg vs Placebo; Hazard Ratio = QAW039 150mg / Placebo; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.54 to 1.22] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Hazard Ratio = QAW039 450mg / Placebo; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.41 to 0.97] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio
Statistical Analysis 3: Comparison: QAW039 150mg vs QAW039 450 mg; Hazard Ratio = QAW039 450mg / QAW039 150mg; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.55 to 1.11] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio

5. Primary Outcome: Number of Participants With Treatment Emergent AEs Leading to Discontinuation From Study Treatment up to Week 52 - Cox Regression Model
Description: Adverse events leading to study treatment discontinuation starting on or after the day of the first intake of study drug in this study and until the day of last intake of study drug +7 days (30 days in the case of a serious AE) were classified as treatment emergent AEs leading to study treatment discontinuation. For this Outcome Measure, AE up to week 52 are reported.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 1081 | 1077 | 359
Participants | 26 | 33 | 9
Statistical Analysis 1: Comparison: QAW039 150mg vs Placebo; Hazard Ratio = QAW039 150mg / Placebo; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.47 to 2.23] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Hazard Ratio = QAW039 450mg / Placebo; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.59 to 2.64] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio
Statistical Analysis 3: Comparison: QAW039 150mg vs QAW039 450 mg; Hazard Ratio = QAW039 450mg / QAW039 150mg; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.70 to 2.10] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio

6. Primary Outcome: Number of Participants With Treatment Emergent AEs Leading to Discontinuation From Study Treatment up to Week 156 - Cox Regression Model
Description: Adverse events leading to study treatment discontinuation starting on or after the day of the first intake of study drug in this study and until the day of last intake of study drug +7 days (30 days in the case of a serious AE) were classified as treatment emergent AEs leading to study treatment discontinuation
Time Frame: 156 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 1081 | 1077 | 359
Participants | 30 | 37 | 9
Statistical Analysis 1: Comparison: QAW039 150mg vs Placebo; Hazard Ratio = QAW039 150mg / Placebo; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.56 to 2.56] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Hazard Ratio = QAW039 450mg / Placebo; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.67 to 2.95] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio
Statistical Analysis 3: Comparison: QAW039 150mg vs QAW039 450 mg; Hazard Ratio = QAW039 450mg / QAW039 150mg; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.70 to 1.96] — A hazard ratio < 1 favors the treatment group in the numerator of the ratio

7. Secondary Outcome: Number of Patients With at Least One Treatment Emergent AE by Primary System Organ Class up to Week 52 - Logistic Regression Model
Description: The number of patients per patient year of follow-up having a treatment emergent adverse event, categorized by system organ class. Treatment emergent adverse events are defined as an AEs starting on or after the day of the first intake of study drug in this study and until the day of last intake of study drug +7 days (30 days in the case of a serious AE)
Time Frame: 52 weeks
Population: Safety analysis set (SAF): included all patients who received at least one dose of study drug during this study. Patients were analyzed according to the treatment they received during this study. Only patients with data for all terms in the Logistic regression model were included
Measure: Count of Participants; unit: Participants
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 1081 | 1077 | 359
Participants
  Number of patients with at least one AE | 675 | 654 | 237
  Blood and lymphatic system disorders | 21 | 10 | 5
  Cardiac disorders | 11 | 26 | 7
  Congenital, familial and genetic disorders | 1 | 3 | 0
  Ear and labyrinth disorders | 16 | 9 | 8
  Endocrine disorders | 2 | 6 | 0
  Eye disorders | 13 | 11 | 9
  Gastrointestinal disorders | 88 | 86 | 32
  General disorders & administration site conditions | 38 | 33 | 7
  Hepatobiliary disorders | 9 | 17 | 7
  Immune system disorders | 11 | 10 | 6
  Infections and infestations | 400 | 374 | 145
  Injury, poisoning and procedural complications | 67 | 52 | 23
  Investigations | 79 | 85 | 20
  Metabolism and nutrition disorders | 53 | 50 | 21
  Musculoskeletal and connective tissue disorders | 91 | 84 | 24
  Neoplasms benign, malignant and unspecified | 13 | 9 | 3
  Nervous system disorders | 67 | 73 | 29
  Product issues | 1 | 0 | 0
  Psychiatric disorders | 18 | 15 | 9
  Renal and urinary disorders | 33 | 41 | 8
  Reproductive system and breast disorders | 14 | 9 | 4
  Respiratory, thoracic and mediastinal disorders | 308 | 304 | 135
  Skin and subcutaneous tissue disorders | 38 | 39 | 13
  Social circumstances | 1 | 1 | 3
  Vascular disorders | 39 | 33 | 9
Statistical Analysis 1: Comparison: QAW039 150mg vs Placebo; Statistical Analysis for Number of patients with at least one AE. Hazard Ratio = QAW039 150mg /Placebo; Test type: Superiority; Regression, Logistic; Logistic regression model: logit (proportion) = randomization stratum, treatment, severity of asthma, region as fixed effects; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.626 to 1.047]
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Statistical Analysis for Number of patients with at least one AE. Hazard Ratio = QAW039 450mg /Placebo; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.622 to 1.038]
Statistical Analysis 3: Comparison: QAW039 150mg vs QAW039 450 mg; Statistical Analysis for Number of patients with at least one AE. Hazard Ratio = QAW039 450mg /QAW039 150mg; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.821 to 1.200]

8. Secondary Outcome: Number of Patients With at Least One Treatment Emergent AE by Primary System Organ Class up to Week 156 - Logistic Regression Model
Description: as for outcome 7
Time Frame: 156 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 1081 | 1077 | 359
Participants
  Number of patients with at least one AE | 710 | 682 | 243
  Blood and lymphatic system disorders | 23 | 12 | 5
  Cardiac disorders | 16 | 34 | 7
  Congenital, familial and genetic disorders | 1 | 3 | 1
  Ear and labyrinth disorders | 18 | 13 | 9
  Endocrine disorders | 5 | 7 | 0
  Eye disorders | 16 | 14 | 9
  Gastrointestinal disorders | 101 | 96 | 38
  General disorders & administration site conditions | 43 | 34 | 8
  Hepatobiliary disorders | 10 | 21 | 8
  Immune system disorders | 11 | 11 | 6
  Infections and infestations | 436 | 415 | 151
  Injury, poisoning and procedural complications | 80 | 63 | 28
  Investigations | 90 | 102 | 24
  Metabolism and nutrition disorders | 61 | 60 | 23
  Musculoskeletal and connective tissue disorders | 102 | 92 | 31
  Neoplasms benign, malignant and unspecified | 17 | 11 | 3
  Nervous system disorders | 83 | 77 | 32
  Pregnancy, puerperium and perinatal conditions | 1 | 0 | 0
  Product issues | 1 | 0 | 0
  Psychiatric disorders | 23 | 18 | 9
  Renal and urinary disorders | 36 | 45 | 10
  Reproductive system and breast disorders | 17 | 10 | 4
  Respiratory, thoracic and mediastinal disorders | 336 | 341 | 144
  Skin and subcutaneous tissue disorders | 45 | 45 | 15
  Social circumstances | 1 | 1 | 3
  Vascular disorders | 45 | 40 | 13
Statistical Analysis 1: Comparison: QAW039 150mg vs Placebo; Statistical Analysis for Number of patients with at least one AE. Hazard Ratio = QAW039 150mg /Placebo; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.667 to 1.125]
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Statistical Analysis for Number of patients with at least one AE. Hazard Ratio = QAW039 450mg /Placebo; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.643 to 1.082]
Statistical Analysis 3: Comparison: QAW039 150mg vs QAW039 450 mg; Statistical Analysis for Number of patients with at least one AE. Hazard Ratio = QAW039 450mg /QAW039 150mg; Test type: Superiority; Regression, Logistic; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.794 to 1.167]

9. Secondary Outcome: Number of Treatment Emergent Patient Deaths Due to an Asthma Exacerbation up to Week 52
Description: The number of treatment emergent patient deaths due to an asthma exacerbation. Treatment emergent deaths are defined as deaths resulting from treatment emergent AEs.
Time Frame: 52 weeks
Population: Safety analysis set (SAF): included all patients who received at least one dose of study drug during this study. Patients were analyzed according to the treatment they received during this study.
Measure: Number; unit: Number of deaths
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 1092 | 1084 | 361
Number of deaths | 0 | 0 | 0

10. Secondary Outcome: Number of Treatment Emergent Patient Deaths Due to an Asthma Exacerbation up to Week 156
Description: as for outcome 9
Time Frame: 156 weeks
Population: as for outcome 9
Measure: Number; unit: Number of deaths
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 1092 | 1084 | 361
Number of deaths | 0 | 0 | 0

11. Secondary Outcome: Rate of Treatment Emergent Severe Asthma Exacerbation Episodes Requiring Hospitalizations Per Person Year up to Week 52
Description: Number of treatment emergent severe asthma exacerbation episodes requiring hospitalizations (any visit to the hospital requiring an overnight stay or an emergency room visit greater than 24 hours) per person year of follow-up. Treatment emergent severe asthma exacerbation episodes are defined as episodes occurring on or after the day of the first intake of study drug and until the day of last intake of study drug +7 days (30 days in the case of a serious AE).
  Rate of exacerbations per person year = total number of exacerbations / total number of treatment years
Time Frame: 52 weeks
Population: as for outcome 9
Measure: Number; unit: Hospitalizations per person year
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 1092 | 1084 | 361
Hospitalizations per person year | 0.04 | 0.02 | 0.06

12. Secondary Outcome: Rate of Treatment Emergent Severe Asthma Exacerbation Episodes Requiring Hospitalizations Per Person Year up to Week 156
Description: as for outcome 11
Time Frame: 156 weeks
Population: as for outcome 9
Measure: Number; unit: Hospitalizations per person year
Arm/Group | QAW039 150mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 1092 | 1084 | 361
Hospitalizations per person year | 0.04 | 0.02 | 0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 7 days post treatment (30 days in the case of a serious AE), up to maximum duration of 156 weeks.
Description: Any sign or symptom that occurs during the study treatment plus the 7 days post treatment (30 days in the case of a serious AE).
Groups:
- QAW039 150 mg: QAW039 150 mg
- QAW039 450 mg: QAW039 450 mg
- Placebo: Placebo
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 3/1092 | 1/1084 | 1/361
Serious Adverse Events (participants affected / at risk) | 87/1092 | 64/1084 | 33/361
Other Adverse Events (participants affected / at risk) | 525/1092 | 499/1084 | 190/361
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 150 mg (N=1092) | QAW039 450 mg (N=1084) | Placebo (N=361)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 2 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Fibrous dysplasia of bone (Congenital, familial and genetic disorders) | 1 | 0 | 0
Skeletal dysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 2
Peritoneal cyst (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Hyperplasia (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0
Swelling face (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 0
Eosinophilic granulomatosis with polyangiitis (Immune system disorders) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 3 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1 | 0
Dengue haemorrhagic fever (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 4 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Vaginal abscess (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Exposure to allergen (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Electrocardiogram Q wave abnormal (Investigations) | 0 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain stem haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0
Colloid brain cyst (Nervous system disorders) | 0 | 1 | 0
Dyspraxia (Nervous system disorders) | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 3 | 0 | 2
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Depression (Psychiatric disorders) | 3 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 1
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 30 | 16 | 13
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 150 mg (N=1092) | QAW039 450 mg (N=1084) | Placebo (N=361)
Bronchitis (Infections and infestations) | 75 | 55 | 38
Influenza (Infections and infestations) | 30 | 28 | 9
Nasopharyngitis (Infections and infestations) | 110 | 106 | 36
Pharyngitis (Infections and infestations) | 34 | 22 | 15
Sinusitis (Infections and infestations) | 39 | 28 | 9
Upper respiratory tract infection (Infections and infestations) | 72 | 43 | 25
Upper respiratory tract infection bacterial (Infections and infestations) | 14 | 31 | 12
Urinary tract infection (Infections and infestations) | 23 | 37 | 11
Viral upper respiratory tract infection (Infections and infestations) | 34 | 31 | 9
Blood creatinine increased (Investigations) | 30 | 42 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 11 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 31 | 10
Headache (Nervous system disorders) | 41 | 29 | 24
Asthma (Respiratory, thoracic and mediastinal disorders) | 291 | 275 | 125
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 19 | 28 | 11
Hypertension (Vascular disorders) | 30 | 30 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-03-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03052517/SAP_000.pdf
  • Study Protocol (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT03052517/Prot_001.pdf